CLINICAL TRIAL: NCT02644902
Title: Effectiveness of Technology Assisted Cascade Training and Supervision of Community Health Workers in Delivering Thinking Healthy Program for Perinatal Depression in a Post-conflict Area of Pakistan- Protocol of a Randomized Controlled Trial
Brief Title: Technology Assisted Cascade Training and Supervision of Community Health Workers for Thinking Healthy Programme
Acronym: THP-TACTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Human Development Research Foundation, Pakistan (Other)
Collaborators: Duke University (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCC-THP-TACTS-2015
Record Dates: First submitted 2015-12-28; First posted 2016-01-01 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Maternal Depression
Keywords: Avatar assisted cascade training and supervision; maternal depression; postconflict; THP

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Technology Arm (Experimental): 5 days training of health workers in THP through avatar assisted cascade training and supervision
  Interventions: Other: Avatar assisted cascade training
- Specialist Arm (Active Comparator): 5 days training and supervision of health workers in THP by specialists
  Interventions: Other: Specialist led training in THP

INTERVENTIONS:
Other: Avatar assisted cascade training — Training of health workers in THP through tablets including avatar characters , and cascaded supervision model.
  Arms: Technology Arm
Other: Specialist led training in THP — Training and supervision of lady health workers by specialists as in original THP
  Arms: Specialist Arm

SUMMARY:
The Thinking Healthy Program is evidence based psychological intervention, delivered by non-specialists, with proven impact on maternal depression. A major challenge in the scale-up of this intervention, especially where health systems are weak, is providing quality training and supervision at scale. Women living in post-conflict areas are at a higher risk of depression than the general population.The key innovation proposed is the development and evaluation of a technology-assisted cascade training and supervision system to assist scale-up of the Thinking Healthy Programme in a post conflict area of Pakistan.

DETAILED DESCRIPTION:
The Thinking Healthy Program (THP) is a cognitive behaviour therapy (CBT)-based intervention for maternal depression, delivered by non-specialists.In a recent meta-analysis commissioned by the WHO, THP was shown to have a large effect and has been adopted by the WHO for global dissemination through its mhGAP programme. A major challenge in the scaling up of this evidence-based intervention is the provision of training and supervision at scale, especially in post-conflict areas with weak health systems. The investigators aim to meet this challenge by providing technology based solutions to training and supervision. Building on the organization's previous work in this area, investigators aim to develop Avatar-assisted cascade training and supervision system that includes: (a) a interactive voice response system for phone based assessment to screen depression in the community; (b) a Tablet-based manual , using special characters or avatars allowing standardized training to be delivered without the need for a specialist trainer; and (c) a cascade training model whereby specialists supervise, from distance, the community health worker program supervisors, who in turn, supervise the community health workers (CHW) as part of their normal routine.

The Lady Health Worker (LHW) Programme covers 85% of Pakistan's rural population through 115,000 LHWs . If this study is able to provide a technological solution to the training and supervision of health workers, they have the potential to provide treatment to an estimated 5 million women in rural Pakistan with maternal depression.

Investigators intend conducting the study in District Swat affected by multiple humanitarian crises in recent years. Swat has a population of 1,257,602 persons, 86% of whom live in rural areas with the average household size of 8.8 persons with a low female literacy. The resurgence of the Taliban movement in the Swat Valley of Pakistan since 2004, and the military operations in 2009 and the displacement of residents created a humanitarian crisis in the area. The devastating floods of 2010 put thousands of people out of their homes, and caused destruction to houses, roads, schools and health facilities.The health infrastructure of a post conflict zone like Swat is particularly fragile with the health workers under threat of being attacked, limiting their mobility. Mental health impacts of conflict are often severe and may not be depicted in the national statistics.

ELIGIBILITY:
Inclusion Criteria:

* Lady health workers currently working in Swat district

Exclusion Criteria:

* Physically unwell, lady health workers on leave

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Competency of health workers in THP skills measured using ENact assessment tool | Immediately after intervention
  The competency of health workers in the two arms will be measured using ENact assessment tool.

SECONDARY OUTCOMES:
Cost of intervention | 3 months after intervention
  Cost of intervention and comparative arm will be assessed from data collected during the trial and analyzed after 3 months.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zafar S, Sikander S, Hamdani SU, Atif N, Akhtar P, Nazir H, Maselko J, Rahman A. The effectiveness of Technology-assisted Cascade Training and Supervision of community health workers in delivering the Thinking Healthy Program for perinatal depression in a post-conflict area of Pakistan - study protocol for a randomized controlled trial. Trials. 2016 Apr 6;17:188. doi: 10.1186/s13063-016-1308-2. PMID 27048477